CLINICAL TRIAL: NCT01221103
Title: Phase I/II Trial of Dexamethasone, Ofatumumab and Bendamustine [Treanda] (DOT) as First-line Treatment of Mantle-cell Lymphoma (MCL) in the Elderly
Brief Title: Dexamethasone, Ofatumumab and Bendamustine (DOT) First-line in Mantle-cell Lymphoma(MCL)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southern Europe New Drug Organization (Other)
Collaborators: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT5909
Record Dates: First submitted 2010-10-13; First posted 2010-10-14 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-09

CONDITIONS: Lymphoma, Mantle-Cell
Keywords: Dexamethasone; Ofatumumab; Bendamustine; Lymphoma, Mantle-Cell; Non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin | interventions — ofatumumab; Bendamustine Hydrochloride

ARMS (1):
- DOT (Experimental): Combination of dexamethasone, ofatumumab and bendamustine
  Interventions: Drug: Combination of dexamethasone, ofatumumab and bendamustine

INTERVENTIONS:
Drug: Combination of dexamethasone, ofatumumab and bendamustine — * Ofatumumab (liquid concentrate for infusion in glass vials) infused iv on day 1 at 300 mg during the first cycle, followed by infusions of 1000 mg on day 1 of each subsequent cycle
  * Bendamustine (powder dissolved in sterile water) infused iv over 30-60 minutes at the dose of 120 mg/m2 (days 2,3 every 21 days) or 120 mg/m2(days 2,3 every 28) or 90 mg/m2 (days 2,3 every 28 days) depending on toxicity
  * Dexamethasone administered i.v. at 40 mg (days 1,2,3,4)
  Other Names: Ofatumumab (HuMax-CD20; ARZERRA); Bendamustine (Treanda; Ribomustin)

SUMMARY:
The rationale for this study design is based on the fact that the maximum tolerated dose (MTD) of single-agent ofatumumab and bendamustine have been previously determined. The choice of the doses for the combination is based on the investigators unpublished clinical experience, as well as inferred from extensive experimental data on the use of other monoclonal antibodies in combination chemotherapy in lymphoma patients. The starting dose of the 2 main component drugs is the MTD of each drug as single agent.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60 years.
2. ECOG Performance Status 0-1.
3. Life expectancy of at least 6 months.
4. Histological diagnosis of MCL (morphology, CD5+/CD20+ /CD23-, t(11:14) and/or cyclin D1 overexpression).
5. Disease requiring treatment (patients with bone marrow only disease, who are candidates for a watch-and-wait approach, will be excluded)
6. Adequate bone marrow, liver and renal function, unless the abnormality is related to the tumor and is unlikely to affect the safety of bendamustine and ofatumumab use. Adequate marrow and organ function will be assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

   * Hemoglobin ≥ 9.0 g/dL
   * Absolute neutrophil count (ANC) ≥ 1000/µl
   * Platelet count ≥ 75000/µl
   * Total bilirubin ≤ 1.5 times the ULN
   * AST and ALT ≤ 2.5 x ULN
   * Alkaline phosphatase ≤ 4 x ULN
   * Serum creatinine ≤ 2.5 x ULN
7. PT-INR/PTT < 1.5 x ULN [Patients who are being therapeutically anticoagulated with agent such as coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists]
8. Written informed consent.

Exclusion Criteria:

1. Previous treatment for mantle-cell lymphoma (MCL)
2. Chronic or current infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis and active Hepatitis C.
3. Other past or current malignancy. Subjects who have been free of malignancy for at least 5 years, or have a history of completely resected non-melanoma skin cancer, or successfully treated in situ carcinoma are eligible.
4. Clinically significant cardiac disease including unstable angina, acute myocardial infarction within 6 months prior to Visit 1, congestive heart failure, and arrhythmia requiring therapy, with the exception of extra systoles or minor conduction abnormalities
5. History of significant cerebrovascular disease or event with significant symptoms or sequelae
6. Glucocorticoid use, unless given in doses ≤ 100 mg/day hydrocortisone (or equivalent dose of other glucocorticoid) for <7 days for exacerbations other than CLL (e.g., asthma)
7. Known HIV positive
8. Subjects who have current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment).
9. Positive serology for Hepatitis B (HB) defined as a positive test for HBsAg. In addition, if negative for HBsAg but HBcAb positive and HBsAb negative, a HB DNA test will be performed and if positive the subject will be excluded. Note: If HBcAb positive and HBsAb positive, which is indicative of a past infection, the subject can be included.
10. Positive serology for hepatitis C (HC) defined by positive test for HCAb, in which case reflexively perform a HC RIBA immunoblot assay on the same sample to confirm the result.
11. Treatment with any known non-marketed drug substance or experimental therapy within 5 terminal half lives or 4 weeks prior to Visit 1, whichever is longer or currently participating in any other interventional clinical study
12. Known or suspected inability to comply with study protocol
13. History of organ allograft
14. Patients with evidence or history of bleeding diathesis.
15. Patients undergoing renal dialysis.
16. Substance abuse, medical psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
17. Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-04 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Adverse events (Phase I) | 60 days after last dose of investigational drug
  Incidence, severity, and attribution of treatment-emergent AEs
Complete Response rate (Phase II) | 24 months
  Response determined according to the revised response criteria for malignant lymphoma (Cheson, JCO 2008)

SECONDARY OUTCOMES:
Duration of response (Phase II) | At the screening, cycle 4 (12 weeks) , cycle 6 (18 weeks), 1 year Follow-up
  Duration estimated from the first confirmed tumor regression to the disease progression.
Serial peripheral blood CD34+ cell counts | Cycles 1 (3 weeks), 4 (12 weeks) and 6 (18 weeks)
Molecular analysis of CD34+ cells | cycle 4 (12 weeks) or cycle 6 (18 weeks for inadequate harvests after cycle 4)
Serial molecular analysis of peripheral blood cells | Cycles 1 (3 weeks), 4 (12 weeks) and 6 (18 weeks)
  Serial molecular analysis by PCR
Ability to harvest ≥ 7 x106 CD34+ cells/kg | Cycle 4 (12 weeks) or cycle 6 (18 weeks for inadequate harvests after cycle 4)
Presence of tumor cells in the peripheral blood | Cycle 1 (3 weeks), 4 (12 weeks) and 6 (18 weeks)
  Monitored by morphology, immunophenotype and PCR

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro M. Gianni, MD, Study Chair — Istituto Nazionale Tumori Milano
Locations (2):
- Italy (2):
  - Fondazione IRCCS Istituto Nazionale Tumori, Milan
  - Ospedali Bianchi - Melacrino - Morelli, Reggio Calabria